CLINICAL TRIAL: NCT06320340
Title: The Effectiveness of Neuromuscular Electrical Stimulation Applied Simultaneously to Exercise on Pain, Range of Motion, Muscle Endurance, Fear of Movement and Disability in Chronic Neck Pain
Brief Title: Effectiveness of NMES on Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aybike Senel, PT, MSc, Research Assistant, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07032024
Record Dates: First submitted 2024-03-09; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Chronic Neck Pain
Keywords: cervical spine; exercise; neck pain; neuromuscular electrical stimulation
MeSH Terms: conditions — Motor Activity; Neck Pain | interventions — Exercise; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator)
  Interventions: Other: Exercise
- Group II (Experimental)
  Interventions: Other: Exercise; Other: Electrotherapy

INTERVENTIONS:
Other: Exercise — the patients were performed following five exercises for 20 minutes of treatment session two days a week for the 8 weeks.: (1) the swan-dive vol. I, (2) the swan-dive vol II., (3) breast stroke preparation vol. I, (4) breast stroke preparation vol. II, and (5) swimming vol. II. All the exercises were repeated for the 10 times in a session. Before the exercises, patients were taught and instructed about the five key elements (lateral expansion, centralization, positioning the chest, the shoulder girdle, and the head) of clinical pilates that they should pay attention to while performing the exercises. In addition, verbal and tactile feedbacks were given to patients during all the treatment sessions to maintain the good posture and to perform exercises properly.
Other: Electrotherapy — Two channels of four-channelled Compex SP Fit-3 (MediCompex SA in Geneva, Switzerland) was used to apply NMES (120 mA, 400 μs, 150 Hz) on lower trapezius and serratus anterior muscles for 20 minutes during exercise.
  Arms: Group II

SUMMARY:
The aim of this randomized-controlled study was to determine the effectiveness of neuromuscular electrical stimulation (NMES) applied simultaneously to exercise on pain, static endurance of cervical deep flexor muscles, fear of movement and disability in chronic neck pain. The participants were randomly assigned to one group which in only five clinical pilates exercises were performed (Group I) or the other group which NMES was applied on lower trapezius and serratus anterior muscles while the same exercises were performing (Group II).

DETAILED DESCRIPTION:
The aim of randomized-controlled study was to determine the effectiveness of neuromuscular electrical stimulation (NMES) applied simultaneously to exercise on pain, static endurance of cervical deep flexor muscles, fear of movement and disability in chronic neck pain. This study, including adults with chronic neck pain aged between 18-65 years, was conducted in laboratory of xxx University from March 2021 to May 2021. The participants were randomly assigned to one group which in only five clinical pilates exercises were performed (Group I) or the other group which NMES was applied on lower trapezius and serratus anterior muscles while the same exercises were performing (Group II). Both groups received 20 minutes of treatment session two days a week for the 8 weeks. The pain intensity, range of motion (ROM), static endurance of cervical deep flexor muscles, fear of movement, and neck disability were assessed with Visual Analogue (VAS), universal goniometer, The Deep Neck Flexor (DNF) Endurance Test, Tampa Scale of Kinesiophobia (TSK) and Neck Disability Index (NDI), respectively. All the assessments were performed twice as before and end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* (1) being aged from 18 to 65 years old,
* (2) having neck pain shows mechanical nature longer than 3 months, and
* (3) getting a score of at least 10 from Neck Disability Index.

Exclusion Criteria:

* (1) having a surgery on neck and shoulder regions,
* (2) having a neurological symptom, and
* (3) did not complete the process of the assessment and intervention of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Neck disability | baseline (first assessment)
  The Neck Disability Index consisted 10 questions investigating the pain intensity and difficulty in lifting, reading, concentration, working, sleeping and recreational activities. Each question is scoring from 0 to 5 and higher score means greater disability.
Neck disability | at the end of the invervention program (8 weeks after from baseline)
  The Neck Disability Index consisted 10 questions investigating the pain intensity and difficulty in lifting, reading, concentration, working, sleeping and recreational activities. Each question is scoring from 0 to 5 and higher score means greater disability.

SECONDARY OUTCOMES:
Pain intensity | baseline (first assessment)
  The neck pain intensity of the participants were assessed with VAS which is a widely used pain assessments in the musculoskeletal disorders. The participants were asked to rate their pain intensity with a mark on a 10 cm line, which starts with "0-no pain" and ends with "10-unbearable pain". The distance of the mark to the 0 point was measured with a ruler and the pain intensity was recorded as cm.
Pain intensity | at the end of the invervention program (8 weeks after from baseline)
  The neck pain intensity of the participants were assessed with VAS which is a widely used pain assessments in the musculoskeletal disorders. The participants were asked to rate their pain intensity with a mark on a 10 cm line, which starts with "0-no pain" and ends with "10-unbearable pain". The distance of the mark to the 0 point was measured with a ruler and the pain intensity was recorded as cm.
Range of Motion | baseline (first assessment)
  Cervical ROM in all six directions (flexion-extension, lateral flexion, and rotation) were assessed with universal goniometer. Universal goniometer were shown to have good to excellent intra-rater and inter-rater reliability to assess ROM of cervical spine (10.1093/ptj/71.2.98). The measurement were performed as described in (https://doi.org/10.21315/mjms2021.28.2.9). The measurement of each six directions were repeated three times and means were recorded as degree.
Range of Motion | at the end of the invervention program (8 weeks after from baseline)
  Cervical ROM in all six directions (flexion-extension, lateral flexion, and rotation) were assessed with universal goniometer. Universal goniometer were shown to have good to excellent intra-rater and inter-rater reliability to assess ROM of cervical spine (10.1093/ptj/71.2.98). The measurement were performed as described in (https://doi.org/10.21315/mjms2021.28.2.9). The measurement of each six directions were repeated three times and means were recorded as degree.
Static endurance of cervical deep flexor muscles | baseline (first assessment)
  Deep Neck Flexor ((longus capitis, longus colli, rectus capitis anterior and lateralis) Endurance Test was used to static endurance of cervical deep flexor muscles. The subjects began in a supine, hook-lying position, with the hands resting on the abdomen. Upon request, with the chin in maximally tucked position and maintained isometrically, the subject lifted the head and neck approximately 2.5 cm from resting position The duration of holding the head position properly was timed, and static endurance of the DNF was recorded as second.
Static endurance of cervical deep flexor muscles | at the end of the invervention program (8 weeks after from baseline)
  Deep Neck Flexor ((longus capitis, longus colli, rectus capitis anterior and lateralis) Endurance Test was used to static endurance of cervical deep flexor muscles. The subjects began in a supine, hook-lying position, with the hands resting on the abdomen. Upon request, with the chin in maximally tucked position and maintained isometrically, the subject lifted the head and neck approximately 2.5 cm from resting position The duration of holding the head position properly was timed, and static endurance of the DNF was recorded as second.
Fear of the movement | baseline (first assessment)
  Tampa Scale of Kinesiophobia is a Likert type questionnaire consisted of 17 questions scoring from "1-strongly disagree" to "4-strongly agree". Scoring of questions 4, 8, 12, and 16 are reversed. The higher score means greater fear of movement.
Fear of the movement | at the end of the invervention program (8 weeks after from baseline)
  Tampa Scale of Kinesiophobia is a Likert type questionnaire consisted of 17 questions scoring from "1-strongly disagree" to "4-strongly agree". Scoring of questions 4, 8, 12, and 16 are reversed. The higher score means greater fear of movement.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Aydın University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared on request.